CLINICAL TRIAL: NCT03843320
Title: Impact of SAVR and TAVR on Patient's Activity and Mobility CAPABILITY Study
Brief Title: Impact of SAVR and TAVR on Patient's Activity and Mobility
Acronym: CAPABILITY
Status: Suspended | Type: Observational
Why Stopped: Reassessing study feasibility
Sponsor: University of Padova (Other)
Collaborators: Edwards Lifesciences (Industry); Ospedale San Bortolo di Vicenza (Other); Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Other Study IDs: CAPABILITY
Record Dates: First submitted 2019-01-24; First posted 2019-02-18 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Aortic Valve Stenosis
Keywords: SAVR; TAVR; Physical function; Aortic valve replacement; Wearable devices; Smart watch; Activity tracker
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- SAVR: Patients with aortic stenosis undergoing surgical aortic valve replacement using an approved medical device for this intended use.
  Patients will be enrolled in this group only if the device is one of the following:
  * INSPIRIS RESILIA;
  * EDWARDS INTUITY;
  * Carpentier-Edwards PERIMOUNT Magna-Ease.
  Interventions: Device: INSPIRIS RESILIA; Device: EDWARDS INTUITY; Device: Carpentier-Edwards PERIMOUNT Magna-Ease
- TAVR: Patients with aortic stenosis undergoing transcatheter aortic valve replacement using an approved medical device for this intended use.
  Patients will be enrolled in this group only if the device is one of the following:
  * SAPIEN 3;
  * SAPIEN XT.
  Interventions: Device: SAPIEN 3; Device: SAPIEN XT

INTERVENTIONS:
Device: SAPIEN 3 — Transcatheter aortic valve replacement
  Groups: TAVR
Device: SAPIEN XT — Transcatheter aortic valve replacement
  Groups: TAVR
Device: INSPIRIS RESILIA — Surgical aortic valve replacement
  Groups: SAVR
Device: EDWARDS INTUITY — Surgical aortic valve replacement
  Groups: SAVR
Device: Carpentier-Edwards PERIMOUNT Magna-Ease — Surgical aortic valve replacement
  Groups: SAVR

SUMMARY:
This is an independent, investigator-initiated, prospective multicenter observational study with restricted grant provided by Edwards Lifesciences that aims to describe baseline (preoperative) physical function and to assess and compare 6-month postoperative changes in the physical function of patients undergoing aortic stenosis (AS) treatment with either transcatheter aortic valve replacement (TAVR) or surgical aortic valve replacement (SAVR) implanted with Edwards valve type ("SAPIEN 3" and "SAPIEN XT" for TAVR; "INSPIRIS RESILIA", "EDWARDS INTUITY" and "Carpentier-Edwards PERIMOUNT Magna-Ease" for SAVR).

Secondary objectives of this study are: to evaluate the validity of wearable devices in assessing physical function in such patients and subjects' compliance in wearing the device also after a very long follow-up time up to 12 months; to assess and compare 6-month postoperative changes in Health-Related Quality of Life (HRQoL), sleep quality, cognitive function of patients undergoing AS treatment with either TAVR or SAVR.

Smart watch activity tracker "Vívoactive® HR" devices by "Garmin©" will be used in the study. Devices will be distributed to the patients at time of baseline assessment, along with a Bluetooth-paired smartphone provided with a prepaid data-only SIM-card and study-customised interface. Patients will be asked to wear the device 24 hours a day, 7 days a week, from the baseline assessment to the last follow-up, 12 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Severe native aortic valve stenosis symptomatic for heart failure or angina;
* Indication to isolated TAVR or SAVR given by heart team;
* TAVR through the trans-femoral approach;
* SAVR by any access;
* Implantation of an Edwards valve type (SAPIEN 3 and SAPIEN XT for TAVR; INSPIRIS RESILIA, EDWARDS INTUITY and Carpentier-Edwards PERIMOUNT Magna-Ease for SAVR);
* Signed informed consent.

Exclusion Criteria:

* Use of walking aids;
* Dyskinesia or Parkinson's disease;
* Reduced survival expectancy due to severe co-morbidities (<1 year);
* Lack of any of inclusion criteria.

Ages: 75 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing TAVR or SAVR
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test (6 MWT) at 1 month | 1 month after treatment with TAVR/SAVR
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
6-minute walk test (6 MWT) at 3 months | 3 months after treatment with TAVR/SAVR
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
6-minute walk test (6 MWT) at 6 months | 6 months after treatment with TAVR/SAVR
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.

SECONDARY OUTCOMES:
validity of the device in measuring physical function | 1, 3, 6 and 12 months after treatment with TAVR/SAVR
  Differences of length between device measurements and observer measurements of the 6-minute walk test (6MWT)
patients' compliance with the device | 1, 3, 6 and 12 months after treatment with TAVR/SAVR
  median hours/day ratio of data recorded combined with the median days/month ratio in which the device was actively collecting data; formula is [(h/d)*(d/m)]
Patient's perceived health status assessed by the 36-Item Short Form Survey (SF-36) | 1, 3, 6 and 12 months after treatment with TAVR/SAVR
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health status, consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health.
  The SF-36 Health Survey items and scales were constructed using the Likert method of summated ratings. Answers to each question are scored (some items need to be recoded). These scores are then summed to produce raw scale scores for each health concept which are then transformed to a 0 - 100 scale.
Health related Quality of Life (HRQoL) assessed by the Toronto Aortic Stenosis Quality of Life Questionnaire (TASQ) | 1, 3, 6 and 12 months after treatment with TAVR/SAVR
  The Toronto Aortic Stenosis Quality of Life Questionnaire (TASQ) is a 16-item, patient reported survey of patient health status, consists of sixteen questions with a 7-point Likert scale answer. The score is the sum of the answer and transformed into a 0-100 scale. The lower the score the better quality of life, the higher the score the worst quality of life.
Sleep quality assessed by the Epworth Sleepiness Scale (ESS) | 1, 3, 6 and 12 months after treatment with TAVR/SAVR
  The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness that is measured by use of a very short questionnaire. This can be helpful in diagnosing sleep disorders.
  The questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 to 3 for eight different situations. The scores for the eight questions are added together to obtain a single number (0-24) where the lowest is the better outcome: a number in the 0-9 range is considered to be normal while a number in the 10-24 range indicates that expert medical advice should be sought.
Cognitive function assessed by the Mini Mental State Examination (MMSE) | 1, 3, 6 and 12 months after treatment with TAVR/SAVR
  The Mini Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.
  It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document an individual's response to treatment.
  Administration of the test takes between 5 and 10 minutes and examines functions including registration (repeating named prompts), attention and calculation, recall, language, ability to follow simple commands and orientation.
  Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainment and age

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Tarantini, MD, Principal Investigator — University of Padova
Locations (2):
- Italy (2):
  - Azienda Ospedaliera di Padova, Padua, PD
  - Azienda ULSS n.8 Berica, Vicenza - Ospedale San Bortolo, Vicenza, VI

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Background] van Geldorp MW, Heuvelman HJ, Kappetein AP, Busschbach JJ, Cohen DJ, Takkenberg JJ, Bogers AJ. Quality of life among patients with severe aortic stenosis. Neth Heart J. 2013 Jan;21(1):21-7. doi: 10.1007/s12471-012-0364-9. PMID 23229811
- [Background] Stortecky S, Schmid V, Windecker S, Kadner A, Pilgrim T, Buellesfeld L, Khattab AA, Wenaweser P. Improvement of physical and mental health after transfemoral transcatheter aortic valve implantation. EuroIntervention. 2012 Aug;8(4):437-43. doi: 10.4244/EIJV8I4A69. PMID 22917726
- [Derived] Lorenzoni G, Azzolina D, Fraccaro C, Di Liberti A, D'Onofrio A, Cavalli C, Fabris T, D'Amico G, Cibin G, Nai Fovino L, Ocagli H, Gerosa G, Tarantini G, Gregori D. Using Wearable Devices to Monitor Physical Activity in Patients Undergoing Aortic Valve Replacement: Protocol for a Prospective Observational Study. JMIR Res Protoc. 2020 Nov 12;9(11):e20072. doi: 10.2196/20072. PMID 33180023